CLINICAL TRIAL: NCT06939049
Title: Development of New Methodologies and Innovative Tools for the diagnoSi and Therapeutic Treatment of uMAni Epithelial Tumors
Acronym: SISTEMA
Status: Recruiting | Type: Observational
Sponsor: ASL Lecce (Other Government)
Responsible Party: Principal Investigator, Prisco Piscitelli, Medical Doctor, sub-investigator, ASL Lecce
Other Study IDs: DDG_1039/2017_ASL_LE
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cancer Risk; Breast Cancer Risk; Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Salivary and bloody sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lung cancer cohort
- Breast cancer cohort
- Control cohort
- Multiple cancer cohort (Gastrointestinal, urogenital, brain, haematologic cancer)

SUMMARY:
The main objective of the SISTEMA project is to develop non-invasive diagnostic tests for the detection and quantification in blood of markers of Mesenchymal Epithelial Transition, a mechanism that characterises certain types of cancer such as breast and lung cancer. Cancer is still one of the leading causes of death in Western countries. In 2014, there were an estimated 1,665,540 new cancer cases and 585,720 deaths in the United States alone. The World Health Organisation (WHO) and Eurostat predict 1,323,600 deaths in Europe, a figure slightly down on previous statistics but still underlining the existence and seriousness of the problem. It is no coincidence that cancer is one of the main areas of investment in the European Horizon 2020 programme. In recent years, the hypothesis that the process of carcinogenesis is driven by the activation of a particular panel of genes/proteins that enable cancer cells to acquire malignant characteristics has become increasingly popular. This process goes by the name Epithelial Mesenchymal Transition (EMT) and characterises all human epithelial tumours. This process allows epithelial tumour cells to acquire mesenchymal characteristics giving them stem, invasive, and chemoresistant properties.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects over the age of 18 years with an established clinical picture of breast or lung cancer (including mesothelioma) who have not yet started chemotherapy or biological therapies for the treatment of the neoplastic disease and who have read, understood and signed the study information sheet with attached Informed Consent to Participation, signing the attached consent.

Exclusion Criteria:

* Pregnant female patients of either sex under the age of 18 years, undergoing previous drug therapy with corticosteroids, chemotherapies, immunosuppressants and anticancer drugs, as well as patients with a previous history of other malignancies or in a terminal state (life expectancy less than 4 weeks).

Furthermore, lung cancer patients with conditions that could potentially interfere metabolically with the L-fucose biomarker tested in the specific project arm will be excluded, i.e. lung cancer patients simultaneously suffering from: cirrhosis of the liver, gastric ulcer, diabetes mellitus, periodontitis, as well as subjects under stressful conditions (in which false positivity to the marker due to adrenalin release could occur).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects diagnosed with breast cancer or diagnosed with lung cancer, including mesothelioma.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and realisation of non-invasive systems for the detection and quantification of biomarkers of Mesenchymal Epithelial Transition in blood and salivary samples. | 6 months
Validation of innovative biomarkers for the diagnosis and monitoring of therapeutic efficacy in epithelial-mesenchymal transition tumours, primarily breast and lung cancer.Development and implementation of non-invasive systems for the detection and quant | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asl Lecce, Lecce, LECCE, Italy

IPD SHARING:
Plan to Share IPD: No